CLINICAL TRIAL: NCT06144840
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy, Safety, and Tolerability of MT-7117 in Adults and Adolescents With Erythropoietic Protoporphyria or X-Linked Protoporphyria
Brief Title: INcreased Sun Exposure Without Pain In Research Participants With EPP or XLP
Acronym: INSPIRE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-7117-A-302; jRCT2031230656 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2023-506735-15-00 (EU CTIS Number)
Record Dates: First submitted 2023-11-17; First posted 2023-11-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Erythropoietic Protoporphyria (EPP); X-Linked Protoporphyria (XLP)
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Protoporphyria, Erythropoietic, X-Linked Dominant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT-7117 (Experimental)
  Interventions: Drug: Dersimelagon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dersimelagon — MT-7117
  Arms: MT-7117
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To investigate the efficacy of MT-7117 on time to onset and severity of first prodromal symptoms (burning, tingling, itching, or stinging) associated with sunlight exposure in adults and adolescents with EPP or XLP.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects provided written informed consent to participate. For minor subjects, both minor's assent and parental consent will be required.
2. Male and female subjects with a confirmed diagnosis of EPP or XLP based on medical history.
3. Subjects aged 12 years to 75 years, inclusive, at Screening.
4. Subjects are willing and able to travel to the study sites for all scheduled visits.
5. In the Investigator's opinion, subject can understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements (including travel and receiving direct sunlight exposure as much as possible).
6. Female subjects who are non-lactating and have a negative urine pregnancy test at baseline visit prior to receiving the first dose of study drug.
7. Female subjects of childbearing potential and male subjects with partner of child-bearing potential currently using/willing to use 2 effective methods of contraception.

Additional screening criteria check may apply for qualification.

Exclusion Criteria:

1. History or presence of photodermatoses other than EPP or XLP.
2. Subjects who are unwilling or unable to go outside in sunlight during daylight hours most days (e.g., between 1-hour post-sunrise and 1 hour pre-sunset) during the study.
3. Presence or history of any hepatobiliary disease, including druginduced liver injury at screening, determined as clinically significant by the Investigator after the discussion with the Sponsor Medical Monitor.
4. Subjects with aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≥ 2.0 × upper limit of normal (ULN) or total bilirubin >1.5 × ULN at Screening.
5. History (in the last 2 years) or presence of alcohol abuse, or abuse of illicit drugs in the opinion of the Investigator.
6. History of melanoma.
7. Presence of squamous cell carcinoma, basal cell carcinoma, or other malignant skin lesions. Any suspicious lesions or nevi will be evaluated. If the suspicious lesion or nevi cannot be resolved through biopsy or excision, the subject will be excluded from the study.
8. History or presence of psychiatric disease judged to be clinically significant by the Investigator and which may interfere with the study evaluation and/or safety of the subjects.
9. Presence of clinically significant acute or chronic renal disease or subjects with an estimated glomerular filtration rate (eGFR) <60 mL/min as calculated by the Chronic Kidney DiseaseEpidemiology Collaboration (CKD-EPI) creatinine equation (2021) for adults and by the Schwartz creatinine equation for adolescents (2009). Modification of Diet in Renal Disease can be used for adults per local recommendations.
10. Presence of any clinically significant disease or laboratory abnormality which, in the opinion of the Investigator, can interfere with the study objectives and/or safety of the subjects.
11. Female subjects who are pregnant, lactating, or intending to become pregnant during the study.
12. Treatment with any of the following medications or therapy within each period before Randomization (Visit 2);

    * Afamelanotide within 3 months
    * Phototherapy within 3 months
    * Cimetidine within 4 weeks
    * Antioxidant agents within 4 weeks, at doses which, in the opinion of the Investigator, may affect study endpoints (including but not limited to beta-carotene, cysteine, pyridoxine).
    * Chronic treatment with any scheduled analgesic agents including, but not limited to, opioids and opioid derivatives such as morphine, hydrocodone, oxycodone, fentanyl, or their combination with other unscheduled analgesics or non-steroidal anti-inflammatory drug (Percocet and Vicodin-like prescription drugs) within 4 weeks.

    Note: Acute use of scheduled narcotics more than 3 months prior to randomization are allowed. Non-steroidal anti-inflammatory drug, aspirin for analgesia, or prior temporary use of scheduled agents within 3 months of screening is allowed.
13. Dermatological treatments with any drugs or supplements which, in the opinion of the Investigator, can interfere with the objectives of the study or safety of the subjects at screening, such as, for example, tanning agents.
14. Subjects who participated in any previous MT-7117 clinical studies.
15. Previous treatment with any investigational agent such as bitopertin, within 12 weeks before Screening or 5 half-lives of the investigational product (whichever is longer).
16. Use of sunscreens with zinc oxide. Note: Sunscreens without zinc oxide are allowed, however their use, in frequency, quantity and body surface area should be maintained relatively stable throughout the duration of the study.
17. History of any hypersensitivity to the active ingredient and/or excipients (lactose monohydrate, hydroxypropylcellulose, carmellose calcium, magnesium stearate, hypromellose, titanium dioxide, talc, polyethylene glycol, iron oxide yellow, iron oxide red, and iron oxide black). (EU ONLY)
18. Subjects who are unable to swallow tablets or have diseases significantly affecting the gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.(EU ONLY)
19. History of any hypersensitivity to the active ingredient and/or excipients contained in MT-7117 IMP (lactose monohydrate, hydroxypropyl cellulose, carmellose calcium, magnesium stearate, hypromellose, titanium dioxide, talc, polyethylene glycol, iron oxide yellow, iron oxide red, and iron oxide black). (UK ONLY)

Additional screening criteria check may apply for qualification.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in average daily sunlight exposure time (minutes) to first prodromal symptom (burning, tingling, itching, or stinging) associated with sunlight exposure between 1 hour post-sunrise and 1 hour pre-sunset at Week 16 | Week 16
  The comparison between MT-7117 treatment group and placebo group will be performed.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) at Week 16. | Week 16
  The comparison between MT-7117 treatment group and placebo group will be performed.
Total number of sunlight-induced pain events defined as prodromal symptoms (burning, tingling, itching, or stinging) with pain rating of 1-10 on the Likert scale during the 16-week double-blind treatment period. | Week 16
  The comparison between MT-7117 treatment group and placebo group will be performed.
Total number of sunlight-induced non-prodrome, phototoxic reactions during the 16-week double-blind treatment period. | Week 16
  The comparison between MT-7117 treatment group and placebo group will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (36):
- United States (13):
  - Marvel Clinical Research, LLC, Huntington Beach, California
  - University of California at San Francisco, San Francisco, California
  - University Of Miami School Of Medicine, Center For Liver Diseases, Miami, Florida
  - MGH, Boston, Massachusetts
  - MetroBoston Clinical Partners, LLC, Brighton, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Kansas City Research Institute, Kansas City, Missouri
  - Icahn School of Medicine at Mount Sinai (ISMMS) - The Mount Sinai Hospital (MSH), New York, New York
  - Wake Forest University Baptist Health, Winston-Salem, North Carolina
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Einstein Medical Center (EMC), Philadelphia, Pennsylvania
  - The University of Texas Medical Branch (UTMB), Galveston, Texas
  - University of Washington, Seattle, Washington
- Royal Melbourne Hospital (RMH), Parkville, Victoria, Australia
- University Multi-Profile Hospital for Active Treatment (UMHAT) St. Ivan Rilski - Porphyria Center, Sofia, Bulgaria
- Institute for Clinical and Experimental Medicine - IKEM, Prague, Czechia
- France (4):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Saint - Andre, Bordeaux
  - CHU Nantes, Nantes
  - Hôpital Bichat - Hospital Bichat-Hopitaux Universitaires Paris Nord Val de Seine, Paris
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Louis-Mourier, Paris
- Italy (7):
  - Azienda Ospedaliera Spedali Civili di Brescia-Universita degli Studi Di Brescia, Brescia
  - Azienda Sanitaria Ospedaliera Santa Croce E Carle - Cuneo, Cuneo
  - Ospedalle Galliera, Genova
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico di Milano, Milan
  - U.O.C. Medicina Interna Azienda ospedaliero Universitaria Policlinico di Modena, Modena
  - IFO-San Gallicano IRCCS, Rome
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) Materno-Infantile - Burlo Garofolo - Clinica Pediatrica, Trieste
- Japan (3):
  - Mazda Hospital, Aki-gun, Hiroshima
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Tokyo Saiseikai Central Hospital, Tokyo
- Universitair Medisch Centrum Rotterdam, Rotterdam, Netherlands
- Instytut Hematologii I Transfuzjologii, Warsaw, Poland
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario De Valencia, Valencia
- United Kingdom (2):
  - Southampton General Hospital - University Hospital Southampton NHS Foundation Trust, Southamption, Southamption
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: No